CLINICAL TRIAL: NCT01796821
Title: A Double-Blind, Vehicle Controlled, Randomized, Phase II Study of SR-T100 Gel on External Genital Warts/Condyloma Acuminate (EGWs)
Brief Title: Efficacy and Safety Profiles of SR-T100 Gel on External Genital Warts/Condyloma Acuminate(EGWs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GESRTGWA
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Condyloma Acuminata; Genital Warts; Condylomata Acuminata; Venereal Warts
Keywords: Condyloma acuminata; Genital warts; Condylomata acuminata; Venereal warts
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle gel (Placebo Comparator): vehicle gel is used as a control group. The maximum daily dosage is 3 times of 400+/-100 mg of gel, meaning no more than 1,500 mg of gel. Patients should wash thoroughly their hands, then squeeze until 4 cm of gel is out from the aluminum tube. Apply gel on the lesion warts and on the clinical normal skin on the treated area.
  Interventions: Drug: Vehicle gel
- SR-T100 gel with 1.0 % SM (Active Comparator): SR-T100 contains 1.0% SM. The maximum daily dosage is 3 times of 400+/-100 mg of gel, meaning no more than 1,500 mg of gel. Patients should wash thoroughly their hands, then squeeze until 4 cm of gel is out from the aluminum tube. Apply gel on the lesion warts and on the clinical normal skin on the treated area.
  Interventions: Drug: SR-T100 gel with 1.0 % SM
- SR-T100 gel with 2.3% SM (Active Comparator): SR-T100 contains 2.3% SM. The maximum daily dosage is 3 times of 400+/-100 mg of gel, meaning no more than 1,500 mg of gel. Patients should wash thoroughly their hands, then squeeze until 4 cm of gel is out from the aluminum tube. Apply gel on the lesion warts and on the clinical normal skin on the treated area.
  Interventions: Drug: SR-T100 gel with 2.3% SM

INTERVENTIONS:
Drug: Vehicle gel — Clinical diagnosed lesion site(s): Topical application once daily with occlusive dressing.
  Clinical normal skin on treated area: Topical application thrice daily without occlusive dressing.
  Total application <1,500 mg gel per day.
  Arms: Vehicle gel
Drug: SR-T100 gel with 1.0 % SM — Clinical diagnosed lesion site(s): Topical application once daily with occlusive dressing.
  Clinical normal skin on treated area: Topical application thrice daily without occlusive dressing.
  Total application <1,500 mg gel per day.
  Arms: SR-T100 gel with 1.0 % SM
Drug: SR-T100 gel with 2.3% SM — Clinical diagnosed lesion site(s): Topical application once daily with occlusive dressing.
  Clinical normal skin on treated area: Topical application thrice daily without occlusive dressing.
  Total application <1,500 mg gel per day.
  Arms: SR-T100 gel with 2.3% SM

SUMMARY:
To evaluate the efficacy of SR-T100 gel by observing total clearance rate of treated baseline EGW(s) on the treated area.

DETAILED DESCRIPTION:
A double-blind, randomized,vehicle-controlled, parallel-group, and dose-ranging study to evaluate the efficacy and safety of SR-T100 gel in patients with EGW(s). The primary efficacy endpoint will be defined as the proportion of patients whose baseline EGW(s) on the treated area achieve total clearance. The efficacy of SR-T100 gel in prevention of new EGW(s) occurrence will be evaluated. Distinct to existing medications for EGWs, SR-T100 gel possesses characteristics of high safety and low LSR causality. SR-T100 gel will be administered on EGW lesion(s) for clearance and on the surrounding clinical normal skin for prevention of new EGW(s) occurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; aged ≥ 20 years old.
2. Patients who accept to enter the study by signing written informed consent.
3. Each patient has 1 to 10 clinically diagnosed EGW(s). If patient has only 1 genital wart, the diameter of the genital wart must be no less than 5 mm.
4. Female patients have lesion(s) on labia majora, labia minora, clitoris and/or groin.
5. Male patients have lesion(s) on glans, shaft and/or foreskin.
6. Each patient has at least 1 histologically proved EGW.
7. Patients agree to apply the study medication on "clinical diagnosed lesion(s)" with occlusive dressing(s) once daily for at least 20 hours per day and "clinical normal skin on the treated area" thrice daily without occlusive dressing.
8. Patients allow diagrammed mapping and photography on genital warts. And patients agree to be used of these data as part of the study data package.
9. Patients in good general health condition (performance status ≤ 2 Eastern Cooperative Oncology Group (ECOG)).
10. Female patients with child-bearing potential must take reliable contraception method(s) during the participation of the study.
11. Patients must agree to use effective boundary barrier for birth control and re-infection of EGW

Exclusion Criteria:

1. Patients with peri-anal warts.
2. Male patients with warts on scrotum or perineum.
3. Patients with other genital infections.
4. Patients with internal genital warts (such as urethral, intra-vaginal, cervical, rectal, or intra-anal genital warts).
5. Patients with active systemic infections.
6. Patients with other genital diseases that may confound evaluation and treatment for genital warts.
7. Patients with immuno-compromised medical condition.
8. Patients have received investigational drug prior to 30 days of randomization visit.
9. Patients with cancer or cancer history within 5 years of the randomization visit.
10. Patients have on-going human papilloma virus (HPV) infection other than genital area.
11. Patients with human immunodeficiency virus (HIV), venereal disease research laboratory (VDRL), or treponema pallidum particle agglutination assay (TPHA) positive result.
12. Female patients have high-grade pathology in Papanicolaou smear tests based on Bethesda system.
13. Female patients are pregnant or lactating.
14. Patients have history of allergy or sensitivity to Solanum undatum plant extract, SM, or SR-T100 gel excipients including carbomer, propylene glycol, and triethanolamine.
15. Patients with prohibited pre-medication or procedures shown below:

    1. Physical modalities, such as laser ablation, electrocautery or cryotherapy, for genital warts treatment on treated area within 4 weeks prior to randomization visit.
    2. Topical administered medication for genital warts treatment, such as polyphenon E, podophyllotoxin, imiquimod, or 5-fluorouracil (5-FU), within 12 weeks prior to randomization.
    3. Medications of cytotoxic, immunomodulator (inhaled and topical steroid not on ano-genital areas are not prohibited), systematic antiviral agent in 4 weeks prior to randomization visit.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-08; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Total clearance rate of baseline lesion(s) | 16 weeks

SECONDARY OUTCOMES:
Total clearance rate of all lesion(s) | 16 weeks
Period duration of achieving total clearance of baseline lesion(s) and new lesion(s) | 16 weeks
Partial clearance rate | 16 weeks
New lesion(s) occurrence rate | 16 weeks
Recurrence rate in the 12-week follow-up time | 28 weeks
Recurrence time period | 28 weeks
Safety: evaluate the changes occurring from baseline to EOT visit | 28 weeks
  including PE, vital sign, lab. test, local skin reaction, and adverse event, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kou-Wha Kuo, PhD, Study Director — G&E Herbal Biotechnology Co., LTD; Cheng-Yang Chou, M.D., Principal Investigator — National Cheng Kung University, Tainan, Taiwan
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan